CLINICAL TRIAL: NCT01016197
Title: Surgical Versus Conservative Treatment of Acute Mallet Fingers; a Randomised Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Mid Cheshire Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Mr Philip Holland, Mersey Deanery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PH1
Record Dates: First submitted 2009-11-18; First posted 2009-11-19 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Finger Injury
Keywords: Soft tissue mallet finger
MeSH Terms: conditions — Finger Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conservative (Active Comparator): Four weeks of splinting followed by mobilisation.
  Interventions: Procedure: Mallet splint for 4 weeks
- Surgery (Experimental): Surgical repair of the tendon with a bone anchor followed by four weeks of splinting and then mobilisation.
  Interventions: Procedure: extensor tendon repair

INTERVENTIONS:
Procedure: extensor tendon repair — Surgical repair of extensor tendon with bone anchor and splinting
  Arms: Surgery
Procedure: Mallet splint for 4 weeks — The patient will wear a "mallet splint" for fours weeks and then mobilise their finger.
  Arms: Conservative

SUMMARY:
The investigators are investigating if surgical treatment of injuries to the tendon which straightens the finger tip gives a better functional outcome than treatment with a splint while the tendon heals.

DETAILED DESCRIPTION:
The investigators will randomise patients to receive splinting of their finger while their tendon heals or have surgical intervention. Surgical intervention will entail fixing the tendon with bone anchors and splinting. Conservative treament involves splinting while the tendon heals. We will then monitor the functional outcome of the hand using the DASH questionare over 18 months.

ELIGIBILITY:
Inclusion Criteria:

* soft tissue mallet finger
* acute injury

Exclusion Criteria:

* ASA 3 or above
* Unable to give informed consent
* Infection in digit affected

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
DASH score | up to 18 months

SECONDARY OUTCOMES:
Range of movement at distal interphalyngeal joint. | 3, 6, 12 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Philip Holland, MBChB, MRCS, Principal Investigator — National Health Service, United Kingdom
Locations (1):
- Mid Cheshire NHS Trust, Crewe, United Kingdom